CLINICAL TRIAL: NCT06208462
Title: Neoadjuvant Therapy of HAIC（GEMOX） Combined With Adebrelimab and Lenvatinib for Resectable Intrahepatic Cholangiocarcinoma With High-risk Recurrence Factors：NEO-ERA-01 Study
Brief Title: Neoadjuvant Therapy of HAIC（GEMOX） Combined With Adebrelimab and Lenvatinib for Resectable Intrahepatic Cholangiocarcinoma With High-risk Recurrence Factors
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Collaborators: Jiangsu Hengrui Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NEO-ERA-01
Record Dates: First submitted 2024-01-06; First posted 2024-01-17 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-01

CONDITIONS: Intrahepatic Cholangiocarcinoma
MeSH Terms: conditions — Cholangiocarcinoma | interventions — lenvatinib; Gemcitabine; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Combined treatment group (Experimental): 1. Preoperative treatment 3 weeks is a course of treatment HAIC (GEMOX) chemotherapy
     1. It is performed within one week after the identification of ICC
     2. Day 1 HAIC (GEMOX) Oxaliplatin 85mg/m2 + Gemcitabine 800mg/m2 Adebrelimab: Day 3 Adebrelimab 1200mg i.v. Lenvatinib 2# qd
  2. Evaluation every 2 courses, up to 4 courses.
  3. Liver resection: It is performed within 1 month after preoperative treatment.
  4. Postoperative treatment: Day 1-14 Capecitabine 1200mg B.I.D.
  Interventions: Drug: Adebrelimab; Drug: Lenvatinib; Drug: Gemcitabine; Drug: Oxaliplatin

INTERVENTIONS:
Drug: Adebrelimab — 1200mg，i.v. , q3w
  Other Names: SHR-1316
Drug: Lenvatinib — 8mg,qd
  Other Names: 4-{3-chloro-4-[(cyclopropylcarbamoyl)amino]phenoxy}-7-methoxyquinoline-6-carboxamide
Drug: Gemcitabine — 800 mg/m2，q3w
  Other Names: Difluorodeoxycytidine Hydrochloride
Drug: Oxaliplatin — 85 mg/m2，q3w
  Other Names: Diaminocyclohexane Oxalatoplatinum

SUMMARY:
Clinical Study on the efficacy and safety of HAIC（GEMOX）and Lenvatinib combined with Adebrelimab neoadjuvant therapy for resectable Intrahepatic Cholangiocarcinoma with high-risk recurrence factors.

DETAILED DESCRIPTION:
Intrahepatic cholangiocarcinoma (ICC) accounts for more than 20% of hepatic malignancies and has become the second most common primary liver tumor worldwide. The incidence of ICC is increasing annually, showing a trend to affecting younger individuals. Treatment options for ICC contain surgical resection, perioperative chemotherapy, liver-directed therapies and systemic therapy such as cytotoxic therapy, targeted therapy and immunotherapy. Adjuvant chemotherapy after ICC resection has become the standard for patients with resected ICC based on the BILCAP trial with better mOS (53 months vs. 36 months, p=0.028) and RFS (25.9 months vs. 17.4 months, p=0.0093). The rationale for neoadjuvant chemotherapy for patients with resectable ICC also suggests a potential advantage according to NEO-GAP. While the effectiveness of hepatic artery infusion chemotherapy (HAIC) has been proven in unresectable ICC, its role in resectable ICC is controversial. The TOPAZ-1 trial demonstrated the efficacy of immune checkpoint blockade in ICC. However, it remains to be seen whether combined therapy above is effective in resectable ICC.

Surgical resection remains the mainstay for ICC therapy, but postoperative patients often have a high tumor recurrence rate. The median time of disease-free survival is 18.5 months, and recurrence rate is 60%-65%. Previous research suggests that the prognosis of ICC depends on several risk factors for recurrence consisting of Stage ≥ Ib (AJCC 8th), tumor size > 5cm, multiple tumor lesions in the same lobe, presence of radiographic major vascular invasion, or lymph node involvement, technically resectable. Further investigation is needed to evaluate the effectiveness of the comprehensive treatment system, which includes HAIC (GEMOX), immunotherapy, neoadjuvant therapy, and surgical resection, for ICC with high-risk recurrence factors.

The goal of this clinical trial is to assess the efficacy and safety of HAIC (GEMOX) and Lenvatinib combined with Adebrelimab neoadjuvant therapy for resectable ICC with high-risk recurrence factors. The primary end point is to evaluate the propotion of treatment completion (including neo-adjuvant therapy and surgery), and the second outcome measures include overall survival (OS), objective response rate (ORR), pathological complete response (pCR) and the recurrence free survival (RFS) of patients after treatment. In order to investigate more effective ICC therapies, participants will undergo 2-4 cycles of HAIC (GEMOX) in combination with Lenvatinib and Adebrelimab. Evaluation will be conducted every 2 cycles, and surgery will be performed when qualified. Capecitabine will be administered for 1-14 days after surgery, and regular follow-up will be conducted.

ELIGIBILITY:
Inclusion Criteria:

1. The patient must sign the informed consent;
2. Age 18-75 years old, male and female;
3. ECOG Physical status Score (PS score) 0 or 1;
4. Patients with ICC who have been pathologically diagnosed (histopathological and/or cytological examination) or clinically diagnosed as having high-risk factors;

   Risk factors are defined as follows:

   Stage ≥Ib, single lesion > 5cm, multiple tumor lesions in the same lobe, technically resectable;Vascular invasion, regional lymph node metastasis, technically resectable
5. Patients with untreated and resectable locally advanced ICC who have been assessed by the surgeon as surgically resectable;
6. The functional indicators of vital organs meet the following requirements

   ① Neutrophils ≥1.5*109/L; Platelet ≥80*109/L; Hemoglobin ≥9g/dl; Serum albumin ≥3g/dl;② Thyroid stimulating hormone (TSH) ≤ 1 times the upper limit of normal, T3, T4 in the normal range;③ Bilirubin ≤ 1.5 times the upper limit of normal value; ALT and AST≤ 2 times the upper limit of normal value;④ Serum creatinine ≤ 1.5 times the upper limit of normal value, creatinine clearance ≥60 ml/min;
7. The subject has at least one measurable lesion (according to RECIST1.1);
8. Fertile women: must agree to abstain from sex (abstain from heterosexual intercourse) or use a reliable, effective method of contraception for at least 120 days from the signing of the informed consent until the final administration of the study drug. Serum HCG test must be negative within 72 hours before randomization. And must be non-lactating.A woman is considered fertile if she has menstruated, has not yet reached postmenopausal status (no continuous periods for ≥12 months, no cause other than menopause has been found), and has not undergone sterilization (such as hysterectomy, bilateral tubal ligation, or bilateral oophorectomy).
9. For male subjects whose partner is a fertile woman, they must agree to abstain from sex or use a reliable, effective method of contraception for at least 120 days from the signing of the informed consent until the final administration of the study drug. Male subjects also had to agree not to donate sperm during the same time period. Male subjects with a pregnant partner are required to use condoms and do not need to use other methods of contraception.

Exclusion Criteria:

1. Pathological diagnosis of hepatocellular carcinoma, mixed hepatocellular carcinoma and other non-cholangiocarcinoma malignant tumor components;
2. Prior systemic therapy and tumor-related surgical treatment (biliary drainage allowed);Patients who relapse after surgery, have received PD1 antibody, PDL1 antibody or CTLA4 antibody, Lenvatinib, chemotherapy in the past; participated in other clinical trials 30 days before screening
3. Previous or co-existing malignancies other than adequately treated non-melanin skin cancer, cervical carcinoma in situ and thyroid papillary carcinoma;
4. Active pulmonary tuberculosis infection. Patients with active pulmonary tuberculosis infection within 1 year prior to enrollment; Had a history of active tuberculosis infection more than 1 year before enrollment, had not received formal anti-tuberculosis therapy or had active tuberculosis;
5. Have an active, known, or suspected autoimmune disease. Subjects with hypothyroidism requiring hormone replacement therapy and skin conditions that do not require systemic therapy are eligible;
6. Long-term acceptance of systemic sex hormones (doses equivalent to > 10mg prednisone per day) or any other form of immunosuppressive therapy. Participants using inhaled or topical corticosteroids may be enrolled;
7. Severe cardiopulmonary and renal dysfunction;
8. Have hypertension that is not well controlled by antihypertensive medication (systolic blood pressure ≥140mmHg or diastolic blood pressure ≥90mmHg);
9. Abnormal coagulation function (PT> 14s), have a tendency to bleed or are receiving thrombolytic or anticoagulant therapy;
10. HBV DNA> 2000IU/ml, HCV RNA> 1000 IU/ml;
11. Had clinically significant bleeding symptoms or a clear tendency to appear within 3 months before enrollment;
12. Active infections that require systemic treatment;
13. Human immunodeficiency virus (HIV, HIV1/2 antibodies) positive;
14. Have a history of psychotropic substance abuse, alcohol abuse or drug use;
15. Have a history of drug allergy;
16. Other factors, as determined by the investigator, that may affect the subject's safety or compliance with the test. Such as a serious illness (including mental illness) requiring co-treatment, serious laboratory abnormalities, or other family or social factors.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2024-01-19 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Propotion of treatment completion | one year
  Propotion of treatment completion (including neo-adjuvant therapy and surgery)

SECONDARY OUTCOMES:
Assess safety and tolerability | one year
  Assess safety and tolerability of HAIC（GEMOX）and Lenvatinib combined with Adebrelimab neoadjuvant therapy
OS | one year
  Overall survival (OS)
pCR | one year
  Pathological Complete Response (pCR)
R0 resection rate | one year
  The percentage of patients received R0 resection after HAIC（GEMOX）and Lenvatinib combined with Adebrelimab neoadjuvant therapy
Major pathological response (MPR) | Until the surgery is over
  Major pathological response (MPR) is defined as ≤50% residual viable tumor cells in the resection bed.
PFS | one year
  Progression-free survival (PFS)
Surgical rate | one year
  The surgical rate of patients after HAIC（GEMOX）and Lenvatinib combined with Adebrelimab neoadjuvant therapy
ORR | one year
  Objective Response Rate （ORR）
Event-free survival (EFS) | one year
  Event-free survival (EFS)
Disease control rate (DCR) | one year
  disease control rate (DCR)

CONTACTS AND LOCATIONS:
Overall Officials: Feng Cheng, MD, Study Director — The First Affiliated Hospital with Nanjing Medical University
Locations (3):
- China (3):
  - The First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - West China Hospital, Chengdu, Sichuan
  - Ningbo Medical Center Lihuili Hospital, Ningbo, Zhejiang